CLINICAL TRIAL: NCT00273585
Title: Randomized Controlled Trial of Software-Based Enhancement of Colorectal Cancer Screening Self-Efficacy
Brief Title: Study of Using Computerized Education to Increase Patients' Confidence in Their Ability to Be Screened for Colon Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Davis (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 200412524-2
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2006-09

CONDITIONS: Colorectal Cancer Screening
Keywords: Fecal occult blood testing; Flexible sigmoidoscopy; Colonoscopy; Self-efficacy

INTERVENTIONS:
Device: Personally-tailored educational software program

SUMMARY:
The purpose of this study is to determine whether a newly developed educational software program is effective in increasing patients' confidence in their ability to undergo colon cancer screening. If the software is effective in this regard, the study will also determine if increased confidence to undergo screening leads to more people being screened and to people feeling as though their decision about screening was informed.

DETAILED DESCRIPTION:
Background: Interactive multimedia computer programs (IMCPs) show promise for facilitating informed patient decisions. However, it is unclear whether IMCPs can activate patients by delivering personally tailored information to bolster self-efficacy, a key mediator of health behavior. It is also unclear whether IMCPs might be employed to lessen disparities in care experienced by less educated people by tailoring self-efficacy enhancing information to educational level and compensating for provider biases in communication. Finally, the optimal way to deploy IMPCs in primary care (e.g. before versus following an office visit) remains unclear. Aims/Hypotheses: We will compare changes in colorectal cancer (CRC) screening self-efficacy, intention, uptake, and informed decision making resulting from an IMCP providing personally tailored information (to subject educational level and self-efficacy) intended to boost self-efficacy with changes resulting from a non-tailored control IMCP. We hypothesize both the intervention and control condition will result in increases in CRC screening self-efficacy, but increases will be significantly greater in the intervention group. We also hypothesize both the intervention and control condition will increase CRC screening intention, uptake, and informed decision making, but increases will be greater in the intervention group and will be mediated by self-efficacy enhancement. Methods: Pilot randomized controlled trial (RCT) of 2 groups, comparing a PCN office visit-linked, tailored (to subject self-efficacy) IMCP software program plus mailed reminders versus a non-tailored CRC screening IMCP software program plus mailed reminders (control). Screening methods targeted will be fecal occult blood testing, flexible sigmoidoscopy, colonoscopy, and computed tomographic virtual colonoscopy. Primary outcomes will be CRC screening self-efficacy, intention, uptake, and informed decision making. Implications: Our pilot is powered to detect a significant effect on CRC screening self-efficacy but not other outcomes; however, by conducting it as we would a future and larger RCT, we will determine protocol feasibility. If our hypotheses are confirmed, it would imply cancer screening IMCPs should be focused on enhancing self-efficacy. Since self-efficacy is a mediator of many patient and health care provider behaviors, it would also imply that similar IMCPs could be developed to support a host of patient and professional education efforts.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50
* Able to read and speak English
* Have a telephone and permanent mailing address
* Have adequate vision, hearing, and hand function to utilize a multimedia software program on a laptop computer
* Lack up to date status for CRC screening

Exclusion Criteria:

* Personal history of biopsy-proven colorectal adenoma or CRC
* Personal history of inflammatory bowel disease involving the colon, unless limited to the rectum
* Current symptoms worrisome for colorectal neoplasm (e.g. rectal bleeding, change in stool caliber)
* Colorectal cancer in 1 or more first degree relatives
* Familial adenomatous polyposis

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-08; Study Completion 2006-02

PRIMARY OUTCOMES:
Colorectal cancer screening self-efficacy

SECONDARY OUTCOMES:
Colorectal cancer screening intention
Colorectal cancer screening decisional conflict

CONTACTS AND LOCATIONS:
Overall Officials: Anthony F Jerant, MD, Principal Investigator — Department of Family & Community Medicine, UC Davis School of Medicine
Locations (1):
- Department of Family & Community Medicine, UC Davis School of Medicine, Sacramento, California, United States